CLINICAL TRIAL: NCT00782249
Title: Prospective Randomized Trial Comparing Different Stimulation Paradigms in Patients Treated With Vagus Nerve Stimulation for Refractory Epilepsy
Brief Title: Trial Comparing Different Stimulation Paradigms in Patients Treated With Vagus Nerve Stimulation for Refractory Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005/238
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 (Experimental): Vagus nerve stimulation paradigm #1
  Interventions: Procedure: Vagus nerve stimulation paradigm #1
- 2 (Experimental): Vagus nerve stimulation paradigm #2
  Interventions: Procedure: Vagus nerve stimulation paradigm #2
- 3 (Experimental): Vagus nerve stimulation paradigm #3
  Interventions: Procedure: Vagus nerve stimulation paradigm #3

INTERVENTIONS:
Procedure: Vagus nerve stimulation paradigm #1 — Vagus nerve stimulation parameters #1
  Arms: 1
Procedure: Vagus nerve stimulation paradigm #2 — Vagus nerve stimulation parameters #2
  Arms: 2
Procedure: Vagus nerve stimulation paradigm #3 — Vagus nerve stimulation parameters #3
  Arms: 3

SUMMARY:
Patients with refractory epilepsy who are candidates for a treatment with vagus nerve stimulation will be prospectively randomized into 3 arms with different vagus nerve stimulation paradigms. Vagus nerve stimulation parameters are programmed and adjusted during outpatient clinic visits, within the normal clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* 16 years or older
* At least 1 seizure/month with alteration of consciousness
* Documented seizure diary, at least 3 months prior to implantation (baseline)
* No change in anti-epileptic drugs 1 month before implantation
* At least one or more AEDs

Exclusion Criteria:

* Active cardiac, pulmonary or gastrointestinal disease
* Vagotomy
* Concomitant use of an investigational drug
* Unstable medical condition
* Unstable psychiatric condition

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-09-28 (Actual); Primary Completion 2009-05-18 (Actual); Study Completion 2009-05-18 (Actual)

PRIMARY OUTCOMES:
Efficacy of vagus nerve stimulation: responder rates and mean monthly seizure frequency reduction, mean seizure free interval, seizure severity and seizure type | After 6 and 12 months

SECONDARY OUTCOMES:
VNS-related side effects | After 6 and 12 months
Battery life | After 6 and 12 months
Quality of life: changes in QOLIE 89 score | After 12 months
Mood assessment: changes in Beck depression scale scores | After 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Boon, MD, PhD, Principal Investigator — University Hospital, Ghent; Vijay Thadani, MD, Principal Investigator — Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
Locations (2):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be